CLINICAL TRIAL: NCT05277220
Title: Evaluation of the Recovery of the Sympathetic Block After Spinal Anesthesia by Thermographic Image
Acronym: THERMOSYMPA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOUAZIZ Hervé, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2021-A01606-35
Record Dates: First submitted 2021-12-06; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Spinal Anesthesia
Keywords: recovery of sympathetic block; thermographic image; outpatient surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thermography
  Interventions: Device: Thermal Camera Thermo Malin TC

INTERVENTIONS:
Device: Thermal Camera Thermo Malin TC — Thermo Malin TC thermal camera (also called HIKVISION TP 31B portable thermal camera). Manufacturer of the researched product is HIKVISION.
  This thermal camera is equipped with a thermal detector with a resolution of 160 x 120 elements or an infrared resolution of 19,200 pixels.
  Thermal sensitivity of the Thermo Malin TC thermal imager is 40 milliKelvin (0.04 °C), with a spatial resolution of 5.48 mrad and a field of view of 37.2 x 50 °. Temperature accuracy at one point varies by +/- 0.5 °C. This thermal imager has four color palettes to highlight the desired elements.
  This camera is specially designed for measuring body temperature in a temperature range from +30 to + 45 °C.
  As part of the research, the thermal camera will enable the acquisition and recording of thermographic images at three times of study. These images are then transferred to the operating software for the Thermo Malin Series to process, analyze and make changes to elements of thermographic images.

SUMMARY:
Spinal anesthesia is a locoregional perimedullary anesthesia which consists of temporary interruption of nerve transmission within the subarachnoid space.

This anesthesia is produced, via a lumbar puncture, by injecting a solution of local anesthetics into cerebrospinal fluid.

Spinal anesthesia generates installation of three consecutive blocks: (i) a sympathetic block (vasodilation, increased skin heat in the sleeping area, arterial hypotension); (ii) a sensory block (i.e. a sensory paralysis: no pain or sensations at the incision), the level of which is assessed by the "touch" test and (iii) a motor block (a motor paralysis : immobility of the limb at the incision) measured by the Bromage score.

Spinal anesthesia is a common method of anesthesia in orthopedic surgery of the lower limbs, as demonstrated by field practice at the Surgical Center Emile Gallé (CCEG). This mode of anesthesia is an alternative to general anesthesia, especially because of a higher benefit / risk ratio. Patients at high-risk will be referred preferentially to a spinal anesthesia to prevent complications related to general anesthesia.

If the regulatory conditions are met (formalized expert recommendations 2009), some orthopedic procedures can be performed in the context of day hospitalization. The constraints of day hospitalization involve the use of anesthetic agents or doses compatible with a short duration of action equivalent to the duration of the act of surgery. They must allow a duration of action of maximum 4 hours, a predictable extension of the block at the T10 level (at the sensory level of the umbilicus), a short period of autonomy in ambulation, a rapid recovery from the dysfunction bladder and absence of hemodynamic effects. The return to normal motor function is the sine qua non of fitness for the street.

The discharge from the post-intervention monitoring room of a patient operated on under spinal anesthesia is validated once the recovery of the 3 blocks has been objectified : the motor block (bromage score), the sensory block (touch test) and the sympathetic block ( hemodynamic parameters).

One of the side effects associated with spinal anesthesia is the installation of a sympathetic block causing more or less significant hemodynamic variations. In current practice, its recovery is objectified when the hemodynamic parameters (FC, PNI) postoperatively (measured every 10 minutes) differ by less than 15% from the basic parameters pre-locoregional anesthesia (LRA). This evolution (with a threshold value of 15%) of the hemodynamic parameters constitutes the reference test (Gold Standard) to objectify a recovery of the sympathetic block. In reality, the criteria on which the recovery of the sympathetic block is based are imperfect because side effects (low blood pressure, nausea, vomiting) can be observed when returning to the outpatient surgery sector's, indicating the presence of a residual block.

Data from literature suggest that thermography would be an interesting alternative tool for evaluating the effectiveness of a nerve block after locoregional anesthesia (LRA). Installation of a nerve block is objectified by the change in temperature of the blocked body areas. In fact, the sympathetic block causes vasodilation in these areas and therefore an increase in local temperatures visible on thermography.

Concretely, performed before locoregional anesthesia (LRA), thermography gives a basal body mapping of local temperatures. These are the reference temperatures.

After performing locoregional anesthesia, the sympathetic block sets in and causes vasodilation which is itself responsible for an increase in local temperatures (appearance of warm colors on the body map). Then the return to the initial temperatures (i.e. those observed at the preoperative time) is done gradually as the sympathetic block recovers.

Use of the thermographic method to detect the recovery of sympathetic block after spinal anesthesia has never been evaluated. However, by comparison to these preoperative images, thermography could allow the detection of areas of local temperatures that are still high postoperatively (persistence of hot colors on the body map), while a return to basic local temperatures is expected. (neutral or cool colors).

This could alert to the persistence of a residual sympathetic block, with areas of the body where vasodilation persists despite the return to normal of hemodynamic parameters, and prevent complications in outpatient surgery sector's.

Main research hypothesis of the investigators is that thermographic image evaluation has very good sensitivity for the recovery of sympathetic block after spinal anesthesia compared to the reference method based on hemodynamic parameters. In addition, second research hypothesis of the investigators is that the recovery of the residual sympathetic block evaluated by thermographic image can reduce the occurrence of subsequent adverse events.

DETAILED DESCRIPTION:
Main objective is the following:

To evaluate the performance of thermography to assess the state of total recovery of the sympathetic block after spinal anesthesia, the evolution of hemodynamic parameters constituting the reference examination.

Secondary objectives are:

* Secondary objective 1: In patients with recovery of the sympathetic block objectified by the evolution of the hemodynamic parameters, compare the cumulative incidence of adverse events subsequent to the recovery of the sympathetic block according to the presence or not of a residual block determined by the thermographic evaluation .
* Secondary objective 2: Evaluate the inter-observer agreement for the evaluation of the state of recovery of the block (2h30 after the spinal anesthesia) from the thermographic images.
* Secondary objective 3: Describe nurses' responses to the acceptability survey for the use of thermography.
* Secondary objective 4: Evaluate the diagnostic performance of temperature deltas to assess the state of total recovery of the sympathetic block after spinal anesthesia, the evolution of hemodynamic parameters constituting the reference examination.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received complete information on the organization of the research and has not opposed their participation and the use of their data
* Adult patients,
* ASA score from I to 3 stabilized
* Outpatient orthopedic surgery of the lower limbs scheduled at the CCEG-Regional University Hospital Center of NANCY
* Locoregional anesthesia by spinal anesthesia
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Documented allergy to one of the agents injected intrathecally
* Uncorrected absolute and / or relative hypovolaemia, as well as situations where the hemodynamics are not stabilized (state of shock, cardiac decompensation, etc.)
* Obstructive heart disease (tight mitral stenosis, tight aortic stenosis, obstructive hypertrophic cardiomyopathy)
* Arterial hypertension uncontrolled
* Constrictive pericarditis
* Obliterating arterial disease of the lower limbs
* Raynaud's syndrome
* Localized infection near the puncture site and / or documented systemic infection
* Infection of the lower limbs like erysipelas
* Hemostatic disorder
* Intracranial hypertension
* Neurodegenerative diseases of the spinal cord
* Congenital malformations (spina bifida)
* Surgical emergency
* Multi visceral failure
* Conventional hospitalization
* Persons referred to in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code:
* Pregnant woman, parturient or nursing mother
* Person deprived of liberty by a judicial or administrative decision
* Person unable to express their consent
* Person undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1 of the Public Health Code
* Minor (not emancipated)
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, ASA (American Society of Anesthesiologists) score from I to 3 stabilized, who are going to have lower limb surgery under spinal anesthesia in outpatient surgery
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Performance of thermography in comparison with hemodynamic parameters (gold standard) | Baseline (J0) is the day when the spinal anesthesia is performed, up to 24 hours
  Evaluation of the state of recovery of sympathetic block ("recovered" / "not recovered") from the thermographic images (before spinal anesthesia, 10 min after spinal anesthesia and 2h30 after spinal anesthesia)

SECONDARY OUTCOMES:
Cumulative incidence of each type of complications related to the persistence of a residual sympathetic block in outpatient surgery sector's | Baseline (J0) is the day when the spinal anesthesia is performed, up to 24 hours
  The complications related to the persistence of a residual sympathetic block are: bradycardia, acute retention of urine, postoperative nausea and vomiting, orthostatic hypotension in outpatient surgery sector's.
  The state of total recovery of the block ("recovered" / "not recovered") will be determined by the thermographic evaluation.
State of recovery of the block 2h30 after spinal anesthesia from the evaluation of thermographic images for each assessor | Baseline (J0) is the day when the spinal anesthesia is performed, up to 24 hours
  The state of recovery ("recovered" / "not recovered") from the block to T2 (2h30 after spinal anesthesia) assessed by five evaluators.
  The investigators can thus compare the inter-observer agreement.
Nurses' responses to the satisfaction questionnaire: acceptability survey for nurses at the Emile Gallé Surgical Center in relation to thermography | Baseline (J0) is the day when the spinal anesthesia is performed, up to 24 hours
  The assessment of nurse anesthetists and operating room nurses on the use of thermography through an anonymous questionnaire.
  The questions will relate to their satisfaction ("satisfied" / "not satisfied"), the speed of use ("time-consuming" / "not time consuming"), the ease of use ("easy" / "difficult"), the frequency of malfunction ("not present" / "rare").
Temperature deltas between T1 and T2 | Baseline (J0) is the day when the spinal anesthesia is performed, up to 24 hours
  Sensitivity (%), specificity (%), positive and negative predictive values (%) of temperature deltas (degrees Celsius).
  The temperature delta (degrees Celsius) between T1 and T2, corresponding to the magnitude of the difference between the "maximum" and "minimum" temperatures determined respectively at T1 and T2, will be determined from the evaluation of the thermographic images.

CONTACTS AND LOCATIONS:
Overall Officials: HERVE BOUAZIZ, professor, Principal Investigator — Central Hospital of Nancy (France)

IPD SHARING:
Plan to Share IPD: No